CLINICAL TRIAL: NCT01460615
Title: Cortisone Treatment for the Prevention of Postoperative Pancreatitis and Pancreatitis-induced Complications After Pancreaticoduodenectomy and Distal Pancreatic Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R11009M
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2011-10

CONDITIONS: Postoperative Complications; Postoperative Pancreatitis
Keywords: Postoperative pancreatitis; Postoperative complications; Delayed gastric emptying; Leakage; Fistula; Acinar cell; Risk patient; Pancreaticoduodenectomy; Whipple; Cortisone
MeSH Terms: conditions — Postoperative Complications; Gastroparesis; Fistula | interventions — Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone

SUMMARY:
The purpose of this randomized, placebo-controlled trial is to investigate whether postoperative pancreatitis and other immediate complications after pancreaticoduodenectomy or distal pancreatic resection may be reduced with cortisone treatment. Treatment is administered to high risk patients (defined by high amount of acinar cells in the cut edge of pancreas).

ELIGIBILITY:
Inclusion Criteria:

* Pancreaticoduodenectomy and distal pancreatectomy patients in Tampere University Hospital

Exclusion Criteria:

* Patients with an ongoing cortisone treatment
* Cefuroxime allergy
* Chronic pancreatitis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2011-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Postoperative overall complications of pancreatic resection | within the first 30 days after surgery
  e.g. Postoperative pancreatic fistula, delayed gastric emptying, postpancreatectomy hemorrhage, biliary fistula, wound infection, postoperative pancreatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Laaninen M, Sand J, Nordback I, Vasama K, Laukkarinen J. Perioperative Hydrocortisone Reduces Major Complications After Pancreaticoduodenectomy: A Randomized Controlled Trial. Ann Surg. 2016 Nov;264(5):696-702. doi: 10.1097/SLA.0000000000001883. PMID 27429037